CLINICAL TRIAL: NCT00531622
Title: An Eight-week, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Saredutant 100 mg Once Daily in Combination With Escitalopram 10 mg Once Daily in Patients With Major Depressive Disorder
Brief Title: An Eight-week Study of Saredutant and Escitalopram as Combination Treatment for Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10290; EudraCT 2007-003159-36
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Episode; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — SR 48968; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saredudant/Escitalopram (Experimental): Saredutant 100 mg and Escitalopram 10 mg once daily for a maximum of 8 weeks
  Interventions: Drug: saredutant (SR48968); Drug: escitalopram
- Placebo and Escitalopram (Active Comparator): Placebo for saredutant and Escitalopram 10 mg once daily for a maximum of 8 weeks
  Interventions: Drug: escitalopram; Drug: placebo
- Placebo (Placebo Comparator): Placebo for saredutant and Placebo for Escitalopram once daily for one week during the screening phase and for a maximum of 8 weeks during the active phase
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: saredutant (SR48968) — oral administration, capsules
  Arms: Saredudant/Escitalopram
Drug: escitalopram — oral administration, capsules
  Arms: Placebo and Escitalopram; Saredudant/Escitalopram
Drug: placebo — oral administration, capsules
  Arms: Placebo; Placebo and Escitalopram

SUMMARY:
The main purpose of this study is to evaluate the efficacy of saredutant 100mg once daily in combination with escitalopram 10mg once daily compared to saredutant placebo in combination with escitalopram 10mg once daily in patients with major depressive disorder. This study also includes a double-placebo group (saredutant placebo in combination with escitalopram placebo).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with recurrent Major Depressive Disorder

Exclusion Criteria:

* Symptoms of current depressive episode for less than 30 days or more than 2 years
* Mild depression, as measured by standard clinical research scales
* Significant suicide risk
* Lack of sexual activity (including masturbation)
* Other psychiatric conditions that would obscure the results of the study
* History of failure to respond to antidepressant treatment
* Pregnancy or breast-feeding

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 in Hamilton depression rating scale (HAM-D) total score | Baseline, Day 56
Change from Baseline to Day 56 in the CGI-S Severity of Illness score | Baseline, Day 56

SECONDARY OUTCOMES:
Change from baseline to Day 56 in the Clinical Global Impression (CGI) severity of illness score | Baseline, Day 56
Change from baseline to Day 56 in HAM-D depressed mood item scores. | Baseline, Day 56
Percentage of patients demonstrating a treatment response | Day 56
  response is defined as a reduction of at least 50% in HAM-D total score between baseline and any post-baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Bromma, Sweden